CLINICAL TRIAL: NCT04586660
Title: An Open-label, Multi-center, Phase 4 Study of XGEVA® (Denosumab) in Chinese Adults and Skeletally Mature Adolescents With Giant Cell Tumor of the Bone
Brief Title: Study of XGEVA® (Denosumab) in Chinese Adults and Skeletally Mature Adolescents With Giant Cell Tumor of the Bone
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180119
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Giant Cell Tumor of Bone
Keywords: Giant cell tumor of bone (GCTB); XGEVA®
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgically unsalvageable disease (Experimental): Participants with surgically unsalvageable disease (eg, sacral, spinal Giant cell tumor of bone [GCTB], or multiple lesions including pulmonary metastases).
  Interventions: Drug: XGEVA®
- Surgically salvageable disease (Experimental): Participants with surgically salvageable disease whose planned on-study surgery is associated with severe morbidity (eg, joint resection, limb amputation, or hemipelvectomy).
  Interventions: Drug: XGEVA®

INTERVENTIONS:
Drug: XGEVA® — Participants will receive XGEVA® 120 mg subcutaneously (SC) once every 4 weeks (Q4W) with a loading dose of 120 mg SC on day 8 and day 15.
  Other Names: Denosumab

SUMMARY:
The study aims to evaluate the efficacy of XGEVA® in Chinese participants with giant cell tumor of bone (GCTB).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Chinese male or female adults aged ≥ 18 years or skeletally mature adolescents (ie, radiographic evidence of at least 1 mature long bone [eg, humerus with closed growth epiphyseal plate]) ≥ 12 years of age.
* Skeletally mature adolescents must weigh at least 45 kg.
* Pathologically confirmed giant cell tumor of bone (GCTB) within 1 year before study enrollment (central pathology review).
* Measurable evidence of active disease within 1 year before study enrollment.
* Participants with surgically unsalvageable disease (eg, sacral, spinal GCTB, or multiple lesions including pulmonary metastases) OR participants whose planned surgery includes joint resection, limb amputation, hemipelvectomy or surgical procedure resulting in severe morbidity.
* Eastern Cooperative Oncology Group performance status ([ECOG PS] of ≤ 2).

Exclusion Criteria:

* Known or suspected current diagnosis of underlying malignancy including high-grade sarcoma, osteosarcoma, fibrosarcoma, malignant giant cell sarcoma.
* Known diagnosis of malignancy derived from non-musculoskeletal system within the past 5 years (participants with definitively treated basal cell carcinoma and cervical carcinoma in situ are permitted).
* Known or suspected current diagnosis of brown cell tumor of bone or Paget's disease.
* Known or suspected current diagnosis of non GCTB giant cell-rich tumors.
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw.
* Active dental or jaw condition which requires oral surgery, including tooth extraction.
* Non-healed wound after dental/oral surgery.
* Planned invasive dental procedure for the course of the study.
* Any planned treatment with intravenous (IV) or oral bisphosphonates during the study.
* Currently receiving other GCTB-specific treatment (eg, radiation, chemotherapy, or embolization).
* Current or previous XGEVA treatment
* Concurrent bisphosphonate treatment
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Female participant is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 5 months after the last dose of XGEVA.
* Female participants of childbearing potential unwilling to use 2 highly effective method of contraception or acceptable method of effective contraception during treatment and for an additional 5 months after the last dose of XGEVA.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening by a serum pregnancy test and/or urine pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 5 months after the last dose of XGEVA.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 5 months after the last dose of XGEVA.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 5 months after the last dose of XGEVA.
* Participant has known sensitivity to any of the products to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the participant and investigator's knowledge.
* Unstable systemic disease including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before enrollment.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.
* Participant has any kind of disorder that compromises the ability of the participant to give written informed consent and/or to comply with study procedures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response | Up to 36 months
  Objective tumor response is defined as the percentage of participants with complete response (CR) or partial response (PR) evaluated based on European Organisation for Research and Treatment of Cancer (EORTC) criteria and Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Time to disease progression or recurrence in participants with unsalvageable giant cell tumor of bone (GCTM) (Cohort 1 only) | From baseline until end of treatment, up to a maximum of 36 months
Number of participants with surgically salvageable giant cell tumor of bone (GCTB) after treatment (Cohort 1 only) | Month 36
Time to disease progression or recurrence for participants with complete response (CR) from time of surgery (Cohort 2 only) | From time of surgery until end of treatment, up to a maximum of 36 months
Number of participants who do not require surgery in participants with salvageable giant cell tumor of bone (GCTB) (Cohort 2 only) | Up to 36 months
Number of participants with surgically downstaging in participants with salvageable giant cell tumor of bone (GCTB) (Cohort 2 only) | Up to 36 months
Change from baseline in bone turnover markers (urinary N-telopeptide [uNTX]/creatinine ratio) | Baseline to Month 36
Change from baseline in severity of pain assessed by Brief Pain Inventory - Short Form (BPI-SF) score | Baseline to Month 36
  Pain severity will be assessed using Brief Pain Inventory - Short Form. The minimum score is 0 (no pain) and the maximum score is 10 (worst pain imaginable). The higher the score means a worse outcome of more pain.
Number of participants who experience one or more treatment-emergent adverse events (TEAEs) | Baseline to end of safety follow-up, up to approximately 37 months
Number of participants who experience adverse events of special interest | Baseline to end of safety follow-up, up to approximately 37 months
  Adverse events of special interest include hypocalcemia, hypercalcemia following investigational product discontinuation, atypical femoral fracture, and osteonecrosis of the jaw.
Serum XGEVA concentration levels | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- China (8):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Third Affiliated Hospital Of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Meidical University Cancer Hospital, Harbin, Heilongjiang
  - Tangdu Hospital of Air Force Medical University, Xi'an, Shaanxi
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com